CLINICAL TRIAL: NCT02618837
Title: Downstream Versus Upstream Strategy for the Administration of P2Y12 Receptor Blockers In Non ST Elevated acUte Coronary Syndromes With Initial Invasive Indication
Brief Title: Downstream Versus Upstream Strategy for the Administration of P2Y12 Receptor Blockers
Acronym: DUBIUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DUBIUS - 0015746
Record Dates: First submitted 2015-10-29; First posted 2015-12-01 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Unstable Angina or Non ST Elevated Myocardial Infarction
Keywords: NSTEMI; NSTEACS; prasugrel; ticagrelor; Downstream versus Upstream strategy
MeSH Terms: conditions — Angina, Unstable; Non-ST Elevated Myocardial Infarction

ARMS (2):
- Downstream strategy arm (Active Comparator): downstream administration strategy of P2Y12 receptor blockers (prasugrel or ticagrelor)
  Interventions: Procedure: Downstream strategy
- Upstream strategy arm (Active Comparator): upstream administration strategy (ticagrelor only)
  Interventions: Procedure: Upstream strategy

INTERVENTIONS:
Procedure: Downstream strategy — At diagnosis:
  Subjects receive a loading dose of aspirin (150-300mg). Administration of clopidogrel is allowed only for patients already receiving clopidogrel
  Pre-procedure:
  Until PCI is performed, all subjects will be maintained at a minimum of 75mg of aspirin (Subjects with clopidogrel may be maintained at a minimum of 75mg of clopidogrel)
  Peri- and post-procedure:
  For all the patients undergoing PCI, both the use of unfractioned heparin and of bivalirudin will be allowed at the time of PCI; choice based upon clinical judgement.
  In this case, subject will be randomized in a 1:1 fashion to prasugrel vs ticagrelor
  At the time of PCI, the loading doses required (according to randomization):
  * Ticagrelor 180mg, maintained at 90mg b.i.d. for at least 12 months
  * Prasugrel 60mg, maintained at a minimum of 75mg of aspirin for at least 12 months plus 10mg of prasugrel* daily for at least 12 months
    * If subject is >75 years old or <60 kg, daily dose of prasugrel should be 5mg
  Arms: Downstream strategy arm
Procedure: Upstream strategy — At the time of diagnosis:
  Subjects randomized in this arm must receive a loading dose of aspirin (150-300 mg) and ticagrelor (180 mg) at admission as soon as possible.
  Pre-procedure:
  All subjects will be maintained at a minimum of 90 mg of ticagrelor b.i.d. and a minimum of 75 mg of aspirin, until coronary angiography is performed.
  Peri- and post-procedure:
  For all the patients undergoing PCI, both the use of unfractioned heparin and of bivalirudin will be allowed at the time of PCI; the choice of the anticoagulant at the time of PCI will be based upon clinical judgement.
  All subjects randomized to the upstream strategy arm will be maintained at a minimum of 90 mg of ticagrelor b.i.d. and a minimum of 75 mg of aspirin, for at least 12 months. If the subject develops hypersensitivity or intolerance to ticagrelor, clopidogrel may be used as a substitute at a dose in accordance with standard hospital practice (to be documented in the eCRF).
  Arms: Upstream strategy arm

SUMMARY:
To evaluate the impact on outcomes of the currently accepted antithrombotic strategies based on the administration of newer P2Y12 receptor blockers (prasugrel and ticagrelor) in a population of non ST elevated ACS (NSTEACS) patients with an initial invasive indication.

Furthermore, to evaluate the effects of bivalirudin administration in comparison to standard therapy with unfractioned heparin (plus provisional anti-GPIIbIIIa) in NSTEACSpatients who undergo PCI and will thus receive these potent antiplatelet agents which may theoretically favor the occurrence of bleedings.

A combined measure of efficacy and safety endpoints, the so-called net clinical benefit (NACE), will be considered at early (30 days) and mid term (12 months) follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 85
* Non ST elevated acute coronary syndrome (unstable angina, non ST elevated myocardial infarction), with an onset of symptoms during the previous 24 hours.
* An initial invasive strategy is chosen (the patient is expected to undergo coronary angiography within 72 h from admission).
* Subject is able to start therapy with a new P2Y12 inhibitor (prasugrel or ticagrelor) OR is on a maintenance dose of clopidogrel or ticlopidine and is able to switch to a new P2Y12 inhibitor (prasugrel or ticagrelor).
* Subject is able to verbally confirm understanding of risks and benefits of dual antiplatelet therapy in coronary acute syndromes and he/she or his/her legally authorized representative provides written informed consent prior to any Clinical Investigation related procedure, as approved by the appropriate Ethics Committee.
* Patient agrees to comply with follow-up evaluations.

Exclusion Criteria:

* Known hypersensitivity/contraindication to aspirin, clopidogrel, prasugrel, ticagrelor, heparin or bivalirudin, or sensitivity to contrast media, which can't be adequately pre-medicated.
* Platelet count <100,000 cells/mm³ or >700,000 cells/mm³, or a white blood cell (WBC) count <3,000 cells/mm³ within 7 days prior to index procedure.
* Shock.
* Have severe hepatic impairment defined as Child Pugh Class C.
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 3 years following screening. (Female subjects of child-bearing potential must have a negative pregnancy test done within 28 days prior to enrollment).
* Other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy.
* Subject is belonging to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff or sponsor staff) or subject unable to read or write.
* Currently participating in investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with current trial endpoints. Subject must agree not to participate in any other clinical investigation for a period of three years following the index procedure, including clinical trials of medication and invasive procedures. Questionnaire-based studies, or other studies that are non-invasive and do not require medication are allowed.
* Prior history of hemorrhagic or ischemic stroke, a transient ischemic attack (TIA), or sub-arachnoid hemorrhage.
* History of intracranial neoplasm, arterovenous malformation, or aneurysm.
* Have received fibrinolytic therapy within 48 hours of entry or randomization into the study.
* Have active pathological bleeding or history of bleeding diathesis.
* Have clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding.
* Have had recent surgery (within 4 weeks of entry into the study) or are scheduled to undergo surgery within the next 2 months.
* Have received a loading dose of a thienopyridine (ticlopidine, clopidogrel or prasugrel) or a maintenance dose of prasugrel or Ticlopidine or Ticagrelor within 7 days of entry into the study.
* Are receiving a GPIIb/IIIa inhibitor (eptifibatide, tirofiban, or abciximab).
* Are receiving warfarin or other coumarin derivatives.
* Are receiving or will receive oral anticoagulation or other oral antiplatelet therapy (except aspirin [ASA]) that cannot be safely discontinued within the next 3 months.
* Are receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX2) inhibitors that cannot be discontinued or are anticipated to require >2 weeks of daily treatment with NSAID or COX2 inhibitors during the study.
* Concomitant therapy with a strong cytochrome P-4503A inhibitor or inducer.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2520 (Estimated)
Dates: Start 2015-12-14 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of NACE (Net Adverse Cardiac Events) at 30 days | 30 days
  NACE (Net Adverse Cardiac Events) defined as a composite of: death from vascular causes (death from cardiovascular causes or cerebrovascular causes and any death without another known cause), non fatal MI, or non fatal stroke, BARC type 3, 4 and 5 bleeding.
Incidence of NACE (Net Adverse Cardiac Events) at 12 months | 12 months
  NACE (Net Adverse Cardiac Events) defined as a composite of: death from vascular causes (death from cardiovascular causes or cerebrovascular causes and any death without another known cause), non fatal MI, or non fatal stroke, BARC type 3, 4 and 5 bleeding.

SECONDARY OUTCOMES:
Incidence of single digit and composite of death from vascular causes, MI, stroke, TIA, severe recurrent ischemia, recurrent ischemia, or other arterial thrombotic event. | 30 days, 12 months
Incidence of death from any cause | 30 days, 12 months
Incidence of any stent thrombosis according to the ARC criteria | 30 days, 12 months
Incidence of target vessel revascularization (TVR). | 30 days, 12 months
Incidence of NACE (Net Adverse Cardiac Events) occurred in the period between admission and coronary revascularization | 30 days, 12 months
  NACE (Net Adverse Cardiac Events) occurred in the period between admission and coronary revascularization defined as a composite of: death from vascular causes (death from cardiovascular causes or cerebrovascular causes and any death without another known cause), non fatal MI, or non fatal stroke, BARC type 2, 3, 4 and 5 bleeding,
Incidence of target lesion revascularization (TLR) | 30 days, 12 months
Incidence of compliance to mandated antiplatelet therapy | 30 days, 12 months
Incidence of BARC type 2, 3, 4 and 5 bleeding (single digit and composite). | 30 days, 12 months
Incidence of all TIMI major, major-life-threatening, and minor bleeding | 30 days, 12 months
Incidence of all CABG surgery-related TIMI major, minor, and composite of TIMI major or minor bleeding | 30 days, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Veneto, Italy

REFERENCES:
- [Derived] Tarantini G, Mojoli M, Varbella F, Caporale R, Rigattieri S, Ando G, Cirillo P, Pierini S, Santarelli A, Sganzerla P, De Cesare N, Limbruno U, Lupi A, Ricci R, Cernetti C, Favero L, Saia F, Roncon L, Gasparetto V, Ferlini M, Ronco F, Ferri L, Trabattoni D, Russo A, Guiducci V, Penzo C, Tarantino F, Mauro C, Marchese A, Castiglioni B, La Manna A, Martinato M, Gregori D, Angiolillo DJ, Musumeci G. Downstream or upstream administration of P2Y12 receptor blockers in non-ST elevated acute coronary syndromes: study protocol for a randomized controlled trial. Trials. 2020 Nov 24;21(1):966. doi: 10.1186/s13063-020-04859-1. PMID 33234137
- [Derived] Tarantini G, Mojoli M, Varbella F, Caporale R, Rigattieri S, Ando G, Cirillo P, Pierini S, Santarelli A, Sganzerla P, Cacciavillani L, Babuin L, De Cesare N, Limbruno U, Massoni A, Rognoni A, Pavan D, Belloni F, Cernetti C, Favero L, Saia F, Fovino LN, Masiero G, Roncon L, Gasparetto V, Ferlini M, Ronco F, Rossini R, Canova P, Trabattoni D, Russo A, Guiducci V, Penzo C, Tarantino F, Mauro C, Corrada E, Esposito G, Marchese A, Berti S, Martinato M, Azzolina D, Gregori D, Angiolillo DJ, Musumeci G; DUBIUS Investigators; Italian Society of Interventional Cardiology. Timing of Oral P2Y12 Inhibitor Administration in Patients With Non-ST-Segment Elevation Acute Coronary Syndrome. J Am Coll Cardiol. 2020 Nov 24;76(21):2450-2459. doi: 10.1016/j.jacc.2020.08.053. Epub 2020 Aug 31. PMID 32882390